CLINICAL TRIAL: NCT03632148
Title: In Vitro Evaluation of the Effect of HepaStem in the Coagulation Activity in Blood of Patients With Liver Disease.
Brief Title: Effect of Liver MSCs in Blood of Patients With Liver Disease.
Acronym: CIRRHOTIQUE01
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Stephenne Xavier, Clinical Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2017/23JUI/331
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver MSCs or Adult Derived Human Liver Stem/progenitor Cells (ADHLSCs) infusions are currently being developed as a therapeutic medicinal product for the treatment of different liver defects. Nevertheless, a main concern for clinicians and health authorities is the risk of therapy-induced thrombosis, which has been reported in several patients after intravenous infusion. Previous studies showed in fact that most MSCs express a procoagulant activity. ADHLSCs could be used to treat acute de-compensated cirrhotic patients due to their immunomodulatory and anti-fibrotic effects. However in these patients, disturbances of coagulation and haemostasis are common and result in profound haemostatic alterations that can lead to thrombosis as well as to bleeding complications. The aim of this study is to evaluate the effect of ADHLSCs in cirrhotic blood compared to control blood.

ELIGIBILITY:
Inclusion Criteria:

* acute de-compensated cirrhotic patients

Exclusion Criteria:

* anticoagulant treatment except for prophylactic heparin treatment
* coagulopathy
* thrombosis
* cancer

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: hospitalised cirrhotic patients in hepatology or intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Blood parameters in tubing loop model | 1 day
  We plan to use the tubing loop model to study the interaction between acute-on-chronic liver failure patient's blood and ADHLSCss. The tubing loop model is a whole blood coagulation in vitro model that mimics the blood flow circulation. It consists of loops made of polyvinyl chloride tubing coated with heparin without any release of heparin in blood. This technique can be used to mimic cell infusion in an in vitro model as close as possible to a patient infusion. Blood parameters are studied after 5 and 60min incubation.
Fibrin formation in thrombodynamics | 1 day
  The thrombodynamics analyser system records and analyses spatiotemporal dynamics of formation of a fibrin clot in a platelet poor plasma (PPP) sample. We plan to use this model to study the interaction between acute-on-chronic liver failure patient's plasma and ADHLSCss.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium